CLINICAL TRIAL: NCT01211327
Title: Topical Cyclosporine in the Treatment of Vernal Keratoconjunctivitis in a Rwandan Eye Clinic; a Prospective Randomized Double-masked Clinical Trial
Brief Title: Topical Cyclosporine for Vernal Keratoconjunctivitis (VKC) in Rwanda
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Funds for Research in Ophthalmology (FRO) of Belgium (Unknown); Novartis (Industry)
Responsible Party: Professor dr. Philippe Kestelyn, University Hospital Ghent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UZ Ghent 003
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Vernal Keratoconjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Cyclosporine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine A (Experimental): Cyclosporine A (CsA) 2% eye drops
  Interventions: Drug: Cyclosporine A
- Dexamethasone (Active Comparator): Dexamethasone 0,1% eye drops
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclosporine A — Cyclosporine 2% eye drops
  Arms: Cyclosporine A
Drug: Dexamethasone — Dexamethasone 0,1% eye drops
  Arms: Dexamethasone

SUMMARY:
Vernal keratoconjunctivitis (VKC) is a bilateral, chronic, external ocular inflammatory disease of unknown cause. It is a fairly common disease in hot, dry environments, representing as much as 3% of severe ophthalmic diseases and up to 33% of all eye pathology seen among young patients in eye clinics in Central Africa. Symptoms and signs can persist for years with an important visual morbidity and social impact. Corneal changes (e.g. corneal ulcers) can be sight threatening, occurring in up to 10% of VKC children. Topical steroid therapy remains the current standard treatment, but in developing countries its use often is chronic and not medically supervised, potentially leading to bacterial infections, steroid-induced glaucoma and cataract. Chromoglycate drops have less side effects but lack the power to control a flare-up. Topical cyclosporine has the potential to offer an efficient but safer alternative to steroid drops in the management of VKC in an African setting. Its safety and efficiency in the management of vernal keratoconjunctivitis have been described in several uncontrolled studies and double-blind, placebo-controlled trials, but those studies were relatively small and involved populations outside Africa with predominantly palpebral and mixed forms of VKC. Controversy still remains on the efficiency of cyclosporine in severe forms of allergic conjunctivitis like VKC. We therefore undertake a larger prospective randomized double-masked, standard treatment controlled clinical trial in Central Africa to compare the short-term efficiency of cyclosporine A (CsA) 2% eye drops, solved in olive oil vehicle, with that of steroid drops in predominantly limbal forms of VKC. During 4 weeks the participants will be randomised to either cyclosporine or dexamethasone as attack treatment for VKC. The 4 weeks thereafter all participants will receive chromoglycate drops as maintenance treatment. Additional objectives are to document any difference in rebound phenomenon while on chromoglycate during the maintenance phase between the 2 treatment groups and to evaluate safety and tolerance of the test medication.

ELIGIBILITY:
Inclusion Criteria:

- at least 5 years of age

Exclusion Criteria:

* being pregnant
* suffering from any other infectious or inflammatory ocular pathology
* using topical/ systemic corticosteroids, antihistamines, non-steroidal anti-inflammatory drugs or immunosuppressives 2 weeks prior to the trial
* been treated with steroid injection 6 months prior to the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Difference in score for symptoms and clinical signs between treatment arms | After 4 weeks at the end of 4 weeks test medication
  Differences in scores for symptoms and clinical signs individually and as a composite score between the treatment arms.
  Symptoms are itchiness, tearing, stinging, discharge and photophobia. Signs are subtarsal scarring, limbal cysts, pseudogerontoxon, pseudomembrane, corneal plaque, shield-ulcer, bulbar hyperaemia, limbal pigmentation, punctate keratitis, tarsal plate papillae, corneal astigmatism, limbal follicles, conjunctivalisation of the cornea and trantas dots.

SECONDARY OUTCOMES:
Speed of symptom/sign reduction | At 2 weeks while on test medication and at 8 weeks at the end of a chromoglycate maintenance phase
  To document any difference between the 2 treatment groups in speed of symptom/sign reduction during the attack treatment and in rebound phenomenon while on chromoglycate during the maintenance phase
Safety and tolerance of the test medication | At 2 weeks while on test medication and at 8 weeks at the end of a chromoglycate maintenance phase
  To evaluate safety and tolerance of the test medication.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kesteleyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Kabgayi Hospital, Gitarama/Muhanga, Rwanda

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be